CLINICAL TRIAL: NCT00212238
Title: Enhanced Internet Behavior Therapy for Treating Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R03 DK60058 (completed 2007)
Record Dates: First submitted 2005-09-19; First posted 2005-09-21 (Estimated); Last update posted 2010-03-18 (Estimated); Status verified 2010-03

CONDITIONS: Obesity
Keywords: obesity; weight loss; Internet; cognitive behavior therapy; computer assisted patient care; human therapy evaluation; physical activity; clinical trial; nutrient intake activity; outcomes research; personal log /diary; reinforcer; self care; social support network; weight control; behavioral /social science research tag; clinical research; human subject; questionnaire
MeSH Terms: conditions — Obesity; Weight Loss; Motor Activity; Feeding Behavior

INTERVENTIONS:
Behavioral: internet behavioral weight loss program

SUMMARY:
The purpose of this study is to compare two Internet-based behavioral weight loss programs.

DETAILED DESCRIPTION:
Given the increasing prevalence of obesity and fact that many adults have a strong preference to lose weight without attending weekly treatment meetings, there is need to develop effective alternatives to behavioral lifestyle interventions requiring less face-to-face contact. The Internet offers exciting opportunities to deliver behavior change interventions that minimize face-to-face interaction. We have recently developed and tested an Internet behavioral weight loss program compared with an Internet educational program in a randomized trial and found the behavioral program produced significantly better weight losses (4.1 kg) at 6 months. Our study clearly establishes the potential for using the Internet to deliver alternative treatment programs; however, treatment efficacy research is needed to further develop an Internet approach that will promote longer-term weight loss. The objectives of the proposed study are I) to enhance our Internet program to develop a state of the art Internet Cognitive-Behavior Therapy (I-CBT) program for obesity treatment; and 2) to conduct a randomized trial comparing the enhanced program with a Minimal CBT program also delivered via the Internet. We propose to recruit 100 overweight adults and randomly assign them to Enhanced Internet CBT or Minimal Internet CBT programs. The Minimal I-CBT condition will be given links to weight loss websites, weekly structured cognitive-behavioral lessons for weight loss, weekly prompting, and an on-line bulletin board. The Enhanced I-CBT program will have these same features plus weekly on-line group therapy sessions, computer-aided self-monitoring diaries, and weekly individual e-mail feedback from a therapist. The primary outcome is weight loss from 0-12 months. Secondary outcomes will examine patterns of weight change and changes in waist, diet, physical activity, and social support. The proposed research has significant implications for expanding the audience served by obesity treatment program by using the Internet. This study utilizes an innovative approach and extends our programmatic research on the development of a cognitive-behavioral Internet treatment for obesity.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25 to 40

Exclusion Criteria:

* heart attack, stroke, cancer in the last 5 years, angina, diabetes that is treated with oral agents or insulin (people with type 2 diabetes whose disease is controlled through diet and exercise alone will be considered eligible), orthopedic or joint problems that would prohibit exercise;
* major psychiatric diagnoses and organic brain syndromes;
* pregnant, lactating, less than 6 months post-partum, or plan to become pregnant w/in 12 mos.
* currently taking weight loss medications or lost > 5% of body weight during the past 6 months;
* intend to move to another city within the 12 month study duration;
* have another family member living in the household enrolled in the study
* heart problems, frequent chest pains, or faintness or dizziness

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100
Dates: Start 2003-09; Study Completion 2006-10

PRIMARY OUTCOMES:
weight change from 0 to 12 months

SECONDARY OUTCOMES:
patterns of weight change (0-3, 3-6, 6-12 months)
change in waist circumference
change in physical activity
change in dietary intake
change in social support

CONTACTS AND LOCATIONS:
Overall Officials: Deborah F. Tate, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States